CLINICAL TRIAL: NCT05591482
Title: Postoperative Outcomes of Trans-abdominal Open Surgical Repair of Traumatic Diaphragmatic Hernias in Adults.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: zagazig 15
Record Dates: First submitted 2022-10-16; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Hernia, Diaphragmatic
MeSH Terms: conditions — Hernia, Diaphragmatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mesh repair — mesh repair of diaphragmatic hernia

SUMMARY:
Objective: Evaluation of our management of acute or chronic traumatic diaphragmatic hernia repair with sutures or mesh.

Between January 2014 and January 2019, a retrospective study on 185 patients with acute and chronic traumatic diaphragmatic hernias was carried out at the general surgery department of Zagazig University. Results both during and after surgery were assessed.

DETAILED DESCRIPTION:
Traumatic diaphragmatic hernias are the outcome of 0.8% to 6% of blunt trauma cases and more than 17% of cases involving thoraco-abdominal-penetrating trauma (TDH) . Chronic traumatic diaphragmatic herniation (CTDH) is a condition that can develop as a result of an enlargement of a defect in the diaphragm brought on by a pressure difference between the thoracic cavity and the abdominal cavity . It is possible that the rupture will not heal on its own due to the inherent pressure difference that exists between the thorax and the abdomen as well as the continuous movement of the diaphragm .

Due to the seriousness of the related organs' injuries, traumatic diaphragmatic rupture presents a complex emergency and typically necessitates a high diagnostic suspicion. The herniated structures may strangulate into the thoracic cavity, and the mortality rate may increase considerably if the traumatic diaphragmatic hernia is not identified and treated in the acute phase of the trauma . These patients may not be diagnosed until weeks, months, or even years after the initial traumatic event, and they may present with acute symptoms related to the cardiovascular system and the digestive tract. A high mortality rate is seen in people with CTDH with viscera that have been strangulated.

Despite advancements in diagnostic technologies, 2.7 - 50% of patients still have a misdiagnosis . Early, accurate diagnosis is now more common thanks to greater experience and the emergence of imaging tools, particularly computed tomography (CT).

A limited number of researches describe acute and chronic traumatic diaphragmatic hernias in terms of intraoperative and postoperative outcomes. To examine the intraoperative and postoperative results of patients with traumatic diaphragmatic hernias repaired using either suture repair or mesh repair in terms of morbidity, mortality rate, and incidence of recurrence, the investigators have established a retrospective cohort analysis for the current investigation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old, male or female, and had an acute or chronic traumatic diaphragmatic hernia

Exclusion Criteria:

* Hiatus hernias, congenital hernias, diaphragmatic tears without herniation of abdominal organs, eventration of the diaphragm, hernias on both sides of the diaphragm, and recurrent diaphragmatic hernia after prior repair

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between January 2014 and January 2019, 185 patients with acute and chronic traumatic diaphragmatic hernia underwent a retrospective observational study at the general surgery department of Zagazig University. Patients who were >18 years old, male or female, and had an acute or chronic traumatic diaphragmatic hernia met the inclusion criteria. Hiatus hernias, congenital hernias, diaphragmatic tears without herniation of abdominal organs, eventration of the diaphragm, hernias on both sides of the diaphragm, and recurrent diaphragmatic hernia after prior repair were all excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
recurrent hernia | 3.5 years
  recurrence of diaphragmatic hernia after repair

IPD SHARING:
Plan to Share IPD: Yes